CLINICAL TRIAL: NCT05574569
Title: Effect of Cognitive Behavior Play Therapy and Culturally Adapted Mindfulness-Based Guided Self-Help for Parents of Children With Emotional and Behavioral Problems
Brief Title: Cognitive Behavior Play Therapy and Culturally Adapted Mindfulness-Based Guided Self-Help for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Irfan (Other)
Collaborators: University of Peshawar (Other)
Responsible Party: Sponsor-Investigator, Muhammad Irfan, Professor & Head, Department of Mental Health, Psychiatry and Behavioural Sciences, Peshawar Medical College
Organization: Peshawar Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mindfulness & Play Therapy
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Emotional Problem; Behavior Problem
Keywords: Play therapy; Mindful parenting; Emotional Problems; Behavioral Problems
MeSH Terms: conditions — Mental Disorders; Problem Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Play Therapy (Experimental): Play therapy will be given to the participants.
  Interventions: Behavioral: Group 1: Play Therapy
- Group 2: Mindful Parenting (Experimental): Mindful parenting worksheets will be given to the parents.
  Interventions: Behavioral: Group 2: Mindful Parenting
- Group 3: (Combined Interventions of both Group 1 & 2) (Experimental): Play therapy will be given to children and in addition, culturally adapted mindful parenting worksheets will be given to the parents of children having emotional and behavioral problems.
  Interventions: Behavioral: Group 3: (Combined Interventions of both Group 1 & 2)
- Group 4: Treatment as usual (No Intervention): No intervention will be given to the participants

INTERVENTIONS:
Behavioral: Group 1: Play Therapy — Play therapy will be given to children having emotional and behavioral problems.
  Arms: Group 1: Play Therapy
Behavioral: Group 2: Mindful Parenting — Culturally adapted mindful parenting worksheets will be given to the parents of children having emotional and behavioral problems.
  Arms: Group 2: Mindful Parenting
Behavioral: Group 3: (Combined Interventions of both Group 1 & 2) — Play therapy will be given to children and in addition, culturally adapted mindful parenting worksheets will be given to the parents of children having emotional and behavioral problems.
  Arms: Group 3: (Combined Interventions of both Group 1 & 2)

SUMMARY:
Emotional and behavioral problems not only affect the Child's life but also have long-lasting effects on families and society and few studies have been carried out to assess these problems. During the critical phase of childhood, a child may face many emotional and social pressures that can develop physical, behavioral, social, and academic problems, negatively impacting on child's school performance, social involvement, self-esteem along with other serious mental health issues. There is a relationship between traditional parenting practices (such as parental control, love, and rejection) and emotional problems of children including depression and anxiety but very little is known about the role of mindful parenting. Globally, many studies have been done on the prevalence of emotional and behavioral problems in children, whereas relatively little is known about the prevalence of child mental health problems and related risk factors in Pakistan. One of the treatments that they are using these days to provide the developmentally appropriate and therefore effective intervention that meets the mental health needs of children is Cognitive Behavior Play Therapy and mindful parenting.

DETAILED DESCRIPTION:
There is a high prevalence of emotional and behavioral problems globally and a similar is reported in the children of Pakistan, in a study conducted in Karachi. However, despite the alarming situation created by this problem, there is a need of developing culturally adapted approaches due to differences from western culture, where these therapies have been developed and used first. In this context, this study is planned to find out the effect of Cognitive Behavior Play Therapy and Culturally Adapted Mindfulness-based guided self-help for parents of children with Emotional and Behavioral Problems.

The study will be carried out using mixed methods; quantitative and qualitative. The qualitative part will consist of a structured interview with a minimum of 10-15 parents, and mental health professionals, respectively, using the interview questionnaires. The data will be analyzed by systematic content and question analysis which will identify the emerging themes and categories. The data will then be reorganized into wider themes, codes, and categories and written for guidelines to culturally adapt the guided self-help worksheets for parents of emotional and behavioral problems of children.

The quantitative phase will be an RCT involving approximately 108 students and parents (in each arm) to assess the effectiveness of "Play Therapy" for students having emotional and behavioral problems and "Mindful parenting" for parents of these children having emotional and behavioral problems. All those who fulfill the diagnostic criteria of emotional and behavioral problems and are studying in schools will be included in the study.

The intervention group of the RCT will receive Play Therapy and mindful parenting intervention in addition to the treatment as usual (TAU) while the control group receives TAU. The assessment will be carried out at baseline and at the end of therapy (8 weeks). Strength and difficulty Questionnaire (SDQ) with children, and Bangor mindful parenting scale, emotional regulation scale, parenting styles, and marital satisfaction scale with parents will be used respectively. Schwartz Outcome Scale will be used at the follow-up to measure the outcome.

ELIGIBILITY:
Inclusion Criteria:

For the quantitative part of the study:

1. children having emotional and behavioral problems in the age range of 10 to 13 years
2. Parents of these children with at least 10 years of educational level.

Exclusion Criteria:

1. Children having epilepsy
2. cerebral palsy
3. learning disability

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 432 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Strength and Difficulty Questionnaire | 8 weeks (2 months)
  Change in the score of the Strength and difficulty questionnaire (SDQ) from baseline to end of therapy. Minimum Score = 0 Maximum Score = 40. Normal score 0-15, Borderline score 16-19, Abnormal score 20-40. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The Bangor Mindful Parenting Scale | 8 weeks (2 months)
  Change in the score of The Bangor Mindful Parenting Scale from baseline to end of therapy. Higher scores mean a worse outcome.
Emotion Regulations Questionnaire | 8 weeks (2 months)
  Change in the score of Emotion Regulations Questionnaire from baseline to end of therapy. The greater the use of emotional regulation strategies, the higher the score will be. Higher scores mean a worse outcome.
Parenting Style Questionnaire | 8 weeks (2 months)
  Change in the score of the Parenting style questionnaire from baseline to end of therapy. Higher scores mean a worse outcome.
Kansas Marital Satisfaction Scale | 8 weeks (2 months)
  Change in the score of the Kansas marital satisfaction scale from baseline to end of therapy. The higher scores mean better marital quality

CONTACTS AND LOCATIONS:
Overall Officials: Mifrah R Sethi, MSc, MPhil, Principal Investigator — Peshawar Medical College
Locations (1):
- Prime Foundation/Private Schools, Peshawar, Khyber Pakhtunkhaw, Pakistan

IPD SHARING:
Plan to Share IPD: No